CLINICAL TRIAL: NCT03527381
Title: Nitric Oxide Supplementation to the Extracorporeal Circulation Line as a Method of Nephroprotection in Cardiac Surgery
Brief Title: Nitric Oxide in Cardiopulmonary Bypass for Renal Protection in Cardiac Surgery
Acronym: NephroNO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nikolay Kamenshchikov (Other)
Responsible Party: Sponsor-Investigator, Nikolay Kamenshchikov, Principal Investigator, Physician Anesthesiologist, Tomsk National Research Medical Center of the Russian Academy of Sciences
Organization: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NephroNO
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases; Cardiomyopathies; Acute Kidney Injury
Keywords: Cardiopulmonary Bypass; Nitric Oxide; Kidney Function Tests; Renal Insufficiency; Protective Agents; Coronary Artery Bypass; Cardiac Surgery
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Cardiomyopathies; Acute Kidney Injury; Renal Insufficiency | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Single-center prospective, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trial participants, data analysts, and report writers are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Experimental): Patients of this group receive treatment with exogenous gaseous nitric oxide supplied directly to the oxygenator in the cardiopulmonary bypass circuit during cardiac surgery.
  Interventions: Drug: Nitric Oxide
- Standard CPB (Placebo Comparator): Patients of this group receive sham-treatment without supplying nitric oxide to the cardiopulmonary bypass circuit (Standard CPB) during cardiac surgery. Considering dilution of nitric oxide at a high ratio of 1 to 25,000 in the gas mixture of the cardiopulmonary bypass circuit (CPB), no addition of any inert gas to the CPB circuit is required in sham-treatment group.
  Interventions: Other: Standard CPB

INTERVENTIONS:
Drug: Nitric Oxide — 40 ppm of exogenous gaseous nitric oxide is supplied directly to the oxygenator in the cardiopulmonary bypass circuit during cardiac surgery.
  Arms: Nitric Oxide
Other: Standard CPB — Standard CPB protocol of delivery of air gas mixture to the cardiopulmonary bypass circuit during cardiac surgery.
  Arms: Standard CPB

SUMMARY:
This prospective randomized study evaluates the nephroprotective effects of exogenous nitric oxide delivered to the extracorporeal circulation circuit during cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
The aim of this work is to study nephroprotective effects of nitric oxide (NO) supplementation to the cardiopulmonary bypass (CPB) circuit during cardiac surgery with normothermic CPB in adult patients. The prospective randomized study is performed in the settings of Federal Cardiology Center. A total of 96 adult patients who underwent cardiac surgery with CPB are enrolled in the study. Patients are randomized to two groups: main group receive NO treatment; control group undergoes sham procedure. In the main group, NO is supplied to the CPB line in a dose of 40 ppm throughout the entire CPB period. The primary endpoint is the frequency of acute kidney injury (AKI). The secondary endpoints are urine output during CPB; uNGAL level 4 h after surgery; plasma concentration of free hemoglobin (Hb); concentrations of NO metabolites (nitrite (NO2-) and nitrate (NO3-)) and the total concentration of metabolites of NO (NOx, μM/mL) in blood plasma in the intraoperative period; concentration of proinflammatory (TNF-α, IL-1β, -6, and -8) and anti-inflammatory mediators (IL-1ra, IL-4) in blood plasma in the intraoperative period. Cumulative fluid balance, diuresis, and Lasix doses are assessed within the first 48 h of the postoperative period. The dynamics of serum creatinine is assessed during the first week following the intervention.

ELIGIBILITY:
Inclusion Criteria:

Age above 18 years; planned primary cardiac intervention with cardiopulmonary bypass including coronary artery bypass grafting, valve surgery, and surgical reconstructions of the left ventricle.

Exclusion Criteria:

Preoperative anemia; the intake of nephrotoxic drugs or the use of X-ray contrast within 72 h before surgery; active phase of endocarditis; emergency surgery; chronic kidney disease; hematologic diseases accompanied by hemolysis; complications of the surgery and the early postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-12-25 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury rate measure | 48 hours after surgery
  The presence of acute kidney injury (AKI) is assessed during 48 hours after surgery. AKI is defined as follows: an increase in serum creatinine ≥ 0.3 mg/dL (≥ 26.5 μM/L) during 48 hours after surgery; an increase in serum creatinine by ≥ 1.5 times compared with the initial preoperative level for seven days after intervention; and urine output < 0.5 mL/kg/h for 6 hours during the first 48 h after surgery.

SECONDARY OUTCOMES:
Urine output measure | During cardiopulmonary bypass
  Urine output values (mL/kg/h) are assessed during cardiopulmonary bypass (CPB).
Urine neutrophil gelatinase-associated lipocalin concentration measure (uNGAL) | 4 hours after surgery
  The level of uNGAL (ng/mL) is assessed 4 hours after the surgery.
Free hemoglobin (Hb) concentration measure | 24 hours after surgery
  Plasma concentrations of Hg (g/L) are assessed during intraoperative period: before sternotomy, 5 minutes after aortic clamping, 5 minutes after aortic declamping, at the end of surgery, and 24 hours after surgery.
Nitric oxide metabolite concentration measure | 24 hours after surgery
  Concentrations of NO metabolites (nitrite (NO2-) and nitrate (NO3-)) (μM/mL) and the total concentration of metabolites of NO (NOx) (μM/mL) in blood plasma are assessed in the intraoperative period: before sternotomy, 5 minutes after aortic clamping, 5 minutes after aortic declamping, at the end of surgery, and 24 hours after surgery.
Proinflammatory mediator concentration measure | 24 hours after surgery
  Concentrations of proinflammatory (TNF-α, IL-1β, -6, and -8) (pg/mL) in blood plasma are assessed in the intraoperative period: before sternotomy, at the end of surgery, 6 hours after surgery, and 24 hours after surgery.
Anti-inflammatory mediator concentration measure | 24 hours after surgery
  Concentrations of anti-inflammatory mediators (IL-1ra, IL-4) (pg/mL) in blood plasma are assessed in the intraoperative period: before sternotomy, at the end of surgery, 6 hours after surgery, and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Popov, MD, PhD, Study Director — Tomsk NRMC

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.

REFERENCES:
- [Derived] Kamenshchikov NO, Anfinogenova YJ, Kozlov BN, Svirko YS, Pekarskiy SE, Evtushenko VV, Lugovsky VA, Shipulin VM, Lomivorotov VV, Podoksenov YK. Nitric oxide delivery during cardiopulmonary bypass reduces acute kidney injury: A randomized trial. J Thorac Cardiovasc Surg. 2022 Apr;163(4):1393-1403.e9. doi: 10.1016/j.jtcvs.2020.03.182. Epub 2020 Jun 25. PMID 32718702